CLINICAL TRIAL: NCT03662399
Title: A Single Centre, Cross-over Study to Evaluate the Effect of a Range of Pre-formed Orthoses on Function of the Foot and Leg to Generate Technical Data on How the Individual Insoles Impact Gait, Distribution of Load and Stability in a Healthy Population.
Brief Title: Francis Biomechanics Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reckitt Benckiser Healthcare (UK) Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NPD85301
Record Dates: First submitted 2018-06-06; First posted 2018-09-07 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Healthy Subject
MeSH Terms: interventions — Foot Orthoses

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Insole A (Experimental): Investigational product - Insole A
  Interventions: Device: Insoles
- Insole B (Experimental): Investigational product - Insole B
  Interventions: Device: Insoles
- Insole C (Experimental): Investigational product - Insole C
  Interventions: Device: Insoles
- Insole D (Experimental): Investigational product - Insole D
  Interventions: Device: Insoles
- Insole E (Experimental): Investigational product - Insole E
  Interventions: Device: Insoles
- Insole F (Experimental): Investigational product - Insole F
  Interventions: Device: Insoles
- Insole G (Experimental): Non-Investigational product - Standard shoe
  Interventions: Other: Standard shoe

INTERVENTIONS:
Device: Insoles — Orthotic Insoles
  Arms: Insole A; Insole B; Insole C; Insole D; Insole E; Insole F
Other: Standard shoe — Standard shoe
  Other Names: Non-Investigational product
  Arms: Insole G

SUMMARY:
This study aims to evaluate the effect of a range of pre-formed orthoses on function of the foot and leg to generate technical data on how the individual insoles impact gait, distribution of load and stability in a healthy population.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects between the ages of 18-60 years inclusive.
2. Subjects who are able to give written informed consent.
3. Subjects who are able to understand the study, cooperate with the study procedures and are able to attend all study assessments.
4. Subjects who are willing to wear a t-shirt and shorts during the study assessments.
5. Subjects who are willing and able to stand for a minimum of two hours at a time during the study assessments.
6. Subject with shoe size between 4.5 to 11 (UK) / 37 to 45 (European).
7. Subjects who can achieve the acceptable fit of standard shoes.
8. Subjects who do not have any walking impairments and can walk without distress. This will be determined through walking at a speed of 3-5 kmph for a distance of 30 m.
9. Subjects with a Foot Posture Index (FPI) between 6 and 9 showing mild pronation as determined by the study Investigator or designees.
10. Subjects with a BMI between 18.5 - 24.9 kg/m2.

Exclusion Criteria:

1. Subjects who are pregnant or who have given birth within the last 6 months.
2. Subjects who have a medical condition that could compromise the use of the orthotic insoles (peripheral vascular disease or sensory neuropathy).
3. Subjects that have Leg Length Discrepancy (LLD) of more than 5 mm. This will be determined using the Downings Sign (7), a test which is used to establish actual versus functional LLD. This will be cross-referenced with anatomical land marks.
4. Subjects that use prescribed or self-administrated orthotics to correct biomechanical or other issues.
5. Subject that have received any previous orthotic treatment.
6. Subjects who have a current or previous injury that has prevented their usual activities for more than 3 weeks in the last year.
7. Subjects with history of lower limb or foot surgery, inflammatory disease, neurological disease, diabetes, leg ulceration, skin grafts or any other condition that in the opinion of the Investigator or designees could interfere with the assessments in this study.
8. Subjects having ischemia or poor blood supply to the feet, Charcot Arthropathy, autoimmune disease (e.g. rheumatoid arthritis) and connective tissue disease (e.g. scleroderma).
9. Subjects demonstrating symptoms of macrovascular diseases (e.g. angina, stroke).
10. Individuals suffering from other conditions affecting the feet, such as infectious foot conditions, which in the opinion of the Investigator or designees, would interfere with the generation of data and risk the spread of infection to other subjects through the use of the standard shoe.
11. Individuals with broken/irritated or damaged skin on their feet.
12. Individuals suffering from relevant product allergies or sensitivities.
13. Individuals who have consulted a healthcare professional for a gait related or foot pain issue.
14. Individuals who were previously in another clinical study within the last 3 months prior to screening assessment.
15. Employees who are directly involved with the study at study site.
16. Any partner or first degree relative of anyone that has a role in the study at the CRO/Site/Sponsor.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 40-60% Male and female recruitment
Enrollment: 24 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2018-08-10 (Actual)

PRIMARY OUTCOMES:
In shoe dynamic pressure (shock absorption and loading pattern) Impact on Gait | 2 hours
  Peak pressure (PP)
In shoe dynamic pressure (shock absorption and loading pattern) Impact on Gait | 2 hours
  Pressure time integral (PTI)
In shoe dynamic pressure (shock absorption and loading pattern) Impact on Gait | 2 hours
  Force time integral (FTI)
In shoe dynamic pressure (shock absorption and loading pattern) Impact on Gait | 2 hours
  Contact area (CA)
In shoe dynamic pressure (shock absorption and loading pattern) Impact on Gait | 2 hours
  Time to peak pressure (TPP)
In shoe dynamic pressure (shock absorption and loading pattern) Impact on Gait | 2 hours
  Contact time (CT)
In shoe dynamic pressure (shock absorption and loading pattern) Impact on Gait | 2 hours
  Centre of pressure (balance/stability)
3D gait analysis | 2 hours
  Rearfoot angle at contact
3D gait analysis | 2 hours
  Maximum rearfoot angle
3D gait analysis | 2 hours
  Rearfoot excursion
3D gait analysis | 2 hours
  Rearfoot eversion velocity
3D gait analysis | 2 hours
  Stride Velocity (m/s)
3D gait analysis | 2 hours
  Tibial rotation
3D gait analysis | 2 hours
  Displacement of centre of mass
3D gait analysis | 2 hours
  Hip drop
3D gait analysis | 2 hours
  Thoracic rotation
3D gait analysis | 2 hours
  Hip drop velocity
3D gait analysis | 2 hours
  Thoracic rotation velocity
3D gait analysis | 2 hours
  kinetic data. This includes vertical force, vertical impulse, ankle inversion moment, ankle eversion moment, knee adduction moment, hip adduction moment and hip abduction moment (maximums, measured in BW).

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Kaux, Professor, Principal Investigator — Centre Hospitalier Universitaire de Liège, Avenue de L'Hòpital , Belgium
Locations (1):
- Centre Hospitalier Universitaire de Liège, Avenue de L'Hòpital, Liège, Belgium